CLINICAL TRIAL: NCT01919892
Title: Longitudinal Study on the Neuroprotective and Neurotrophic Effects of Lithium in Bipolar Disorder: Identification of Cellular and Molecular Targets Clinically Relevant
Brief Title: Longitudinal Study on the Neuroprotective and Neurotrophic Effects of Lithium
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Sao Paulo (Other)
Responsible Party: Principal Investigator, Rodrigo Machado Vieira, Professor, University of Sao Paulo
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Lithium001; 09/14891-9 (Other: Fapesp)
Record Dates: First submitted 2013-07-10; First posted 2013-08-09 (Estimated); Last update posted 2013-08-09 (Estimated); Status verified 2013-08

CONDITIONS: Bipolar Disorder; Bipolar Depression
Keywords: predictors of response; bipolar disorder; depression; lithium treatment; biomarkers
MeSH Terms: conditions — Bipolar Disorder; Depression | interventions — Lithium

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Lithium 450-900mg/day (Experimental): An Open-Label, 6-week Pilot Study of Flexible Dose of Lithium in Bipolar Depression: The Effectiveness of Lower Lithium Levels
  Interventions: Drug: Lithium

INTERVENTIONS:
Drug: Lithium

SUMMARY:
Thirty subjects with a DSM-IV (Diagnostic and Statistical Manual, fourth version)diagnosis of BPD during a depressive or hypomanic episode will be divided in two groups according to age and time of illness. All patients will receive lithium (flexible therapeutic dose) for 6 weeks and improvement will be evaluated weekly using depression and mania rating scales; this study also objectives to identify state/trait markers and predictors of response.

DETAILED DESCRIPTION:
Mood disorders are the most prevalent psychiatric, presenting chronic course and high morbidity, affecting 10-15% of population. Diverse structural, functional and biochemical cerebral changes described in the pathophysiology of mood disorders, in special Bipolar Disorder (BPD), have been associated with impairments in neuroprotective mechanisms and cellular resilience. However, the clinical relevance of these pathophysiological findings have been rarely addressed. Meanwhile, lithium has been considered the most used mood stabilizer worldwide, showing significant efficacy in the treatment of manic and depressive episodes, as well as in the prevention of suicide and maintenance. Several studies have demonstrated significant neuroprotective and neurotrophic effects induced by lithium treatment in diverse cellular and molecular targets, but again, few is known about the potential association between these cerebral effects and the its therapeutic clinical efficacy induced by this proof of concept agent. The present project aims to investigate brain levels of lithium using magnetic resonance spectroscopy (7Li-MRS) and its association with different markers of neuronal viability such as n-acetyl-aspartate (using 1-hydrogen-MRS), as well as peripheral markers of mitochondrial, endoplasmic reticulum and neurotrophic factors activity, all highly implicated in the pathophysiology of BD. The investigator has been working in this area in the last ten years, in which the last three and a half in the Lab of Molecular Pathophysiology and Experimental Therapeutics, National Institute of Mental Health (NIMH), National Institutes of Health. The candidate is looking forward to establish appropriate structure to develop a "Research Center for the Study of Neuroplasticity and Neuroprotection in Psychiatric Disorders" in the Institute of Psychiatry, University of Sao Paulo, Brazil. Overall, the study on the neuroplasticity-mediated pathophysiological basis of BPD implicated in the clinical presentation and outcome may shed light on the development of new, improved therapeutics for this and other devastating psychiatric disorders.

ELIGIBILITY:
Inclusion Criteria:

* outpatients
* 18-45 yo
* DSM-IV diagnosis of bipolar disorder (BD-I or BD-II)
* current depressive episode based on the Structured Clinical Interview for the Diagnostic and Statistical Manual for Mental Disorders(SCID-I)
* Hamilton Depression Rating Scale Score (HAM-D) ≥18

Exclusion Criteria

* Medical and psychiatric Comorbidity
* more than 5 years of disease duration
* presence of rapid cycling

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2010-09; Primary Completion 2012-11 (Actual); Study Completion 2012-11 (Actual)

PRIMARY OUTCOMES:
Hamilton Depression Rating Scale (HAM-D) | 6 week

SECONDARY OUTCOMES:
Montgomery Asberg Depression Rating Scale (MADRS) | 6 week

OTHER OUTCOMES:
Young Mania Rating Scale | 6 week
  Evaluation of potential switch process to mania in Bipolar Disorder

CONTACTS AND LOCATIONS:
Overall Officials: Rodrigo Machado-Vieira, MD, PhD, Principal Investigator — Institute and Department of Psychiatry, University of Sao Paulo, Brazil
Locations (1):
- Institute of Psychiatry, University of Sao Paullo, São Paulo, São Paulo, Brazil

REFERENCES:
- [Derived] Zanetti MV, Otaduy MC, de Sousa RT, Gattaz WF, Busatto GF, Leite CC, Machado-Vieira R. Bimodal effect of lithium plasma levels on hippocampal glutamate concentrations in bipolar II depression: a pilot study. Int J Neuropsychopharmacol. 2014 Oct 31;18(6):pyu058. doi: 10.1093/ijnp/pyu058. PMID 25522399